CLINICAL TRIAL: NCT03247790
Title: An Open-Label, Two-Period Study to Evaluate the Pharmacokinetics of Lasmiditan in Migraineurs During Acute Migraine Attacks and During Inter-Ictal Periods
Brief Title: A Study of Lasmiditan in Participants With Migraine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 16854; H8H-MC-LAHC (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-08-10; First posted 2017-08-14 (Actual); Results first posted 2019-12-02 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2018-01

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — lasmiditan

STUDY DESIGN:
Intervention Model Description: Multi-center, open-label study with 2 study periods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lasmiditan (Period 1) (Experimental): 200 mg Lasmiditan tablet given once orally during migraine attack.
  Interventions: Drug: Lasmiditan
- Lasmiditan (Period 2) (Experimental): 200 mg Lasmiditan tablet given once orally during inter-ictal period.
  Interventions: Drug: Lasmiditan

INTERVENTIONS:
Drug: Lasmiditan — Administered orally
  Other Names: LY573144

SUMMARY:
The purpose of this study is to measure how much of the drug gets into the blood stream and how long it takes the body to get rid of it during an acute migraine attack and also during the time between acute migraine attacks.

Information about any side effects that may occur will also be collected.

This study includes two study periods. Each study period requires an overnight stay in the Clinical Research Unit (CRU) for at least one night (and up to three nights), followed by up to two outpatient appointments. This study will last approximately 5-6 weeks (not including screening).

Follow-up is required four to seven days after last dose of investigational drug. Screening is required within 28 days prior to the start of the study.

This study is for research purposes only and is not intended to treat any medical condition.

ELIGIBILITY:
Inclusion Criteria:

* Males or females with history of migraine with or without aura, as defined by International Headache Society (IHS) International Classification of Headache Disorders (ICHD)-3 beta guidelines (1.1 and 1.2) (ICHD-3 beta, Cephalalgia 2013), for at least 1 year, based on medical history
* Have a body mass index (BMI) of 18.0 to 40.0 kilograms per meter squared (kg/m²) inclusive, at the time of screening

Exclusion Criteria:

* Have known allergies to lasmiditan, related compounds, or any components of the formulation of lasmiditan
* Have participated, within the last 30 days, in a clinical study involving an investigational product. If the previous investigational product has a long half-life, 5 half-lives or 30 days (whichever is longer) should have passed
* Have an abnormal blood pressure, defined as systolic blood pressure less than or equal to (≤) 90 or greater than (>) 155 millimeters of mercury (mmHg) or diastolic blood pressure ≤ to 50 or >95 mmHg
* Have clinically significant electrocardiogram (ECG) findings, including a QT interval corrected for heart rate using QT interval corrected for heart rate using Fridericia's formula (QTcF) value >450 milliseconds (ms) (males) or >470 ms (females), clinically significant bradycardia, cardiac block, or bradyarrhythmias
* Have a history of, show evidence of, or are undergoing treatment for significant active neuropsychiatric disease (for example, manic depressive illness, schizophrenia, major depressive disorder)
* Have a history of gastrointestinal surgery, or a history of or current irritable bowel syndrome, mal-absorptive disorders, or other gastrointestinal motility disorders. Appendectomy, splenectomy, and cholecystectomy are considered as acceptable
* Have used or intend to use any migraine prevention treatments (including, but not limited to, propranolol or topiramate) within 30 days prior to dosing and until the follow-up visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - eStudySite, San Diego, California
  - AGA Clinical Trials, Hialeah, Florida
  - Meridien Research Inc., Tampa, Florida

REFERENCES:
- See also: A Study of Lasmiditan in Participants With Migraine — https://www.lillytrialguide.com/en-US/studies/headache/LAHC#?postal=

RESULTS

PARTICIPANT FLOW:
Groups:
- Lasmiditan: Participants were administered a single oral dose of 200 mg lasmiditan tablet on 2 occasions (Day 1 of each period) during a migraine attack (Period 1) and during their inter-ictal period (Period 2).
Period: Period 1: Migraine Attack
Arm/Group | Lasmiditan
Started | 16
Received at Least One Dose of Study Drug | 16
Completed | 16
Not Completed | 0
Period: Period 2: Inter-ictal Period
Arm/Group | Lasmiditan
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study drug.
Arm/Group | Lasmiditan
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.8 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 10
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of Lasmiditan in Each Period
Description: PK: Cmax of Lasmiditan in Each Period.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8,12, 18, 24, 48, and 72h post-dose
Population: All enrolled participants who received at least one dose of study drug and have evaluable pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Lasmiditan (Period 1): Participants were administered a single oral dose of 200 mg Lasmiditan tablet on day 1 during migraine attack.
- Lasmiditan (Period 2): Participants were administered a single oral dose of 200 mg Lasmiditan tablet on day 1 during during inter-ictal period.
Arm/Group | Lasmiditan (Period 1) | Lasmiditan (Period 2)
Number analyzed (Participants) | 16 | 16
nanogram per milliliter (ng/mL) | 233 (47) | 227 (44)

2. Primary Outcome: PK: Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of Lasmiditan in Each Period
Description: PK: AUC(0-∞) of Lasmiditan in Each Period.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8,12, 18, 24, 48, and 72h post-dose
Population: All enrolled participants who received at least one dose of study drug and have evaluable pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Lasmiditan (Period 1) | Lasmiditan (Period 2)
Number analyzed (Participants) | 13 | 14
nanogram*hour per milliliter (ng*h/mL) | 1570 (43) | 1640 (46)

3. Secondary Outcome: PK: Maximum Observed Drug Concentration (Cmax) of Major Lasmiditan Metabolites [M3, M8, M7, (S,R)-M18and (S,S)-M18] in Each Period
Description: PK: Cmax of Major Lasmiditan Metabolites [M3, M8, M7, (S,R)-M18and (S,S)-M18] in Each Period.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 18, 24, 48, and 72h post-dose
Population: All enrolled participants who received at least one dose of study drug and have evaluable pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Lasmiditan (Period 1) | Lasmiditan (Period 2)
Number analyzed (Participants) | 16 | 16
ng/mL
  Metabolite: M3 | 14.5 (54) | 14.8 (41)
  Metabolite: M8 | 319 (34) | 326 (30)
  Metabolite: M7 | 77.2 (52) | 85.9 (42)
  Metabolite: (S,R)-M18 | 57.0 (31) | 59.5 (34)
  Metabolite: (S,S)-M18 | 14.0 (37) | 15.0 (27)

4. Secondary Outcome: PK: Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of Major Lasmiditan Metabolites [M3, M8, M7, (S,R)-M18and (S,S)-M18] in Each Period
Description: PK: AUC(0-∞) of Major Lasmiditan Metabolites [M3, M8, M7, (S,R)-M18and (S,S)-M18] in Each Period.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 18, 24, 48, and 72h post-dose
Population: All enrolled participants who received at least one dose of study drug and have evaluable pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Lasmiditan (Period 1) | Lasmiditan (Period 2)
Number analyzed (Participants) | 16 | 16
ng*h/mL
  Metabolite: M3: number analyzed (Participants) | 14 | 13
  Metabolite: M3 | 68.0 (44) | 77.8 (33)
  Metabolite: M8: number analyzed (Participants) | 14 | 15
  Metabolite: M8 | 6180 (28) | 6380 (27)
  Metabolite: M7: number analyzed (Participants) | 14 | 15
  Metabolite: M7 | 820 (80) | 949 (60)
  Metabolite: (S,R)-M18: number analyzed (Participants) | 13 | 16
  Metabolite: (S,R)-M18 | 1460 (33) | 1570 (34)
  Metabolite: (S,S)-M18: number analyzed (Participants) | 9 | 14
  Metabolite: (S,S)-M18 | 363 (29) | 318 (24)

ADVERSE EVENTS:
Time Frame: Up To 58 Days
Description: All enrolled participants who received at least one dose of study drug and had at least one post-dose safety assessment. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Groups:
- Lasmiditan (Period 2): Participants were administered a single oral dose of 200 mg Lasmiditan tablet on day 1 during inter-ictal period.
Arm/Group | Lasmiditan (Period 1) | Lasmiditan (Period 2)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 16/16 | 12/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Lasmiditan (Period 1) (N=16) | Lasmiditan (Period 2) (N=16)
Photophobia (Eye disorders) | 9 (9) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (8) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Vulvovaginitis (Infections and infestations) | 0/14 (0) | 1/14 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0)
Electrocardiogram T wave abnormal (Investigations) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 5 (6) | 6 (6)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 16 (31) | 4 (5)
Paraesthesia (Nervous system disorders) | 9 (9) | 4 (4)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Phonophobia (Psychiatric disorders) | 4 (4) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 2 (2) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Details of the study and its results shall not be publicized in any form without prior consent of the Sponsor. Such approval is necessary to prevent premature disclosure of trade secrets and other confidential information..

DOCUMENTS (2):
  • Study Protocol (2017-07-13): https://cdn.clinicaltrials.gov/large-docs/90/NCT03247790/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-11): https://cdn.clinicaltrials.gov/large-docs/90/NCT03247790/SAP_001.pdf